CLINICAL TRIAL: NCT00722683
Title: Characterization of Breast Masses Using a New Method of Ultrasound Contrast Agent Imaging in 3D Mapping of Vascular Anomalies
Brief Title: Evaluate Breast Masses Using a New Method of Ultrasound Contrast to Detect Abnormal Blood Flow in Breasts
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jerry LeCarpentier PhD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2001-0184
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer; Breast Abnormalities
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound Imaging (Experimental): Ultrasound Imaging with Contrast
  Interventions: Procedure: Ultrasound Imaging with Contrast

INTERVENTIONS:
Procedure: Ultrasound Imaging with Contrast — An ultrasound contrast agent, Definity, will be administered started through the IV line already in use. The imaging will be performed to map vascular flow.
  The breast will be scanned by a double ultrasound transducer system in a holder over the area of the breast to be biopsied. The machine will be set with different settings and the scan repeated, possibly multiple times.

SUMMARY:
The purpose of this study is to determine if breast imaging with ultrasound can be improved by using 1) a ultrasound attachment with two transducers and 2) a contrast agent. These changes might allow smaller blood vessels to be seen than under the way breast ultrasound is usually performed.

DETAILED DESCRIPTION:
The purpose of this study is to determine if performing ultrasound with an attachment made up of two transducers (rather than just a single transducer) will provide more information about the blood vessels in the breast than the current attachment.

The study will also examine the question of whether use of an ultrasound contrast agent will the scanner to see smaller blood vessels than are detected without the agent.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects who have breast masses and scheduled for core biopsy.

Exclusion Criteria:

* Pregnant or lactating females.
* Females who have heart problems or sensitivity to contrast agents.
* Females who have had previous surgery for breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-04; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry L. LeCarpentier, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No